CLINICAL TRIAL: NCT02897297
Title: Observatoire Brestois Des Néoplasies Myéloprolifératives
Brief Title: Myeloproliferative Neoplastic Diseases Observatory From Brest
Acronym: OBENE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: OBENE
Record Dates: First submitted 2016-08-26; First posted 2016-09-13 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
All patients diagnosed or followed in Brest University Hospital for Philadelphia negative myeloproliferative neoplasms will be included in this observational study.

Myeloproliferative neoplasms recorded included: polycythemia vera, essential Thrombocythemia and Primary Myelofibrosis.

This is a not interventional study. Alive patients need to sign a non-opposition consent form.

Patients will be followed until last news (death, change of reference centre...).

DETAILED DESCRIPTION:
In this retrospective and prospective study, clinical and biological data from diagnosis until last news will be recorded.

Clinical data collected: patients and disease characteristics at the time of the diagnosis, disease and mutational status, cardio-vascular risk factors, history of thrombosis and cancer.

Biological data collected: hemogram and bone marrow results if available. During the follow-up new data will be noted: treatment changes (reasons of change and type of drug), thrombotic events (localization, date and hemogram), phenotypic evolutions (type and date), death (date and etiology).

ELIGIBILITY:
Inclusion Criteria:

* Patients with essentiel thrombocythemia, polycythemia vera or primary myelofibrosis
* Signature of the non-opposition consent form

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for essentiel thrombocythemia, polycythemia vera or primary myelofibrosis
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 10 years
  occurrence of death

SECONDARY OUTCOMES:
Incidence of evolutions | 10 years
  occurrence of transformation into polycythemia vera, secondary myelofibrosis, myelodysplastic syndrome or acute leukemia
Incidence of thromboses | 10 years
  occurrence of arterial or venous thrombotic events

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Ianotto, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delluc A, Lacut K, Pan-Petesch B, Galinat H, Lippert E, Ianotto JC. Statin exposure and thrombosis risk in patients with myeloproliferative neoplasms. Thromb Res. 2018 Jul;167:57-59. doi: 10.1016/j.thromres.2018.05.014. Epub 2018 May 16. No abstract available. PMID 29787944
- [Result] Mollard LM, Chauveau A, Boyer-Perrard F, Douet-Guilbert N, Houot R, Quintin-Roue I, Couturier MA, Dagorne A, Malou M, Le Calloch R, Luycx O, Thepot S, Hunault M, Guillerm G, Berthou C, Ugo V, Lippert E, Ianotto JC. Outcome of Ph negative myeloproliferative neoplasms transforming to accelerated or leukemic phase. Leuk Lymphoma. 2018 Dec;59(12):2812-2820. doi: 10.1080/10428194.2018.1441408. Epub 2018 Apr 4. PMID 29616837
- [Result] Mansier O, Luque Paz D, Ianotto JC, Le Bris Y, Chauveau A, Boyer F, Conejero C, Fitoussi O, Riou J, Adiko D, Touati M, Chauzeix J, Viallard JF, Bene MC, Giraudier S, Ugo V, Lippert E. Clinical and biological characterization of MPN patients harboring two driver mutations, a French intergroup of myeloproliferative neoplasms (FIM) study. Am J Hematol. 2018 Aug;93(4):E84-E86. doi: 10.1002/ajh.25014. Epub 2018 Jan 12. No abstract available. PMID 29266414
- [Result] Le Calloch R, Lacut K, Le Gall-Ianotto C, Nowak E, Abiven M, Tempescul A, Dalbies F, Eveillard JR, Ugo V, Giraudier S, Guillerm G, Lippert E, Berthou C, Ianotto JC. Non-adherence to treatment with cytoreductive and/or antithrombotic drugs is frequent and associated with an increased risk of complications in patients with polycythemia vera or essential thrombocythemia (OUEST study). Haematologica. 2018 Apr;103(4):607-613. doi: 10.3324/haematol.2017.180448. Epub 2017 Dec 15. PMID 29246923
- [Result] Ianotto JC, Chauveau A, Boyer-Perrard F, Gyan E, Laribi K, Cony-Makhoul P, Demory JL, de Renzis B, Dosquet C, Rey J, Roy L, Dupriez B, Knoops L, Legros L, Malou M, Hutin P, Ranta D, Benbrahim O, Ugo V, Lippert E, Kiladjian JJ. Benefits and pitfalls of pegylated interferon-alpha2a therapy in patients with myeloproliferative neoplasm-associated myelofibrosis: a French Intergroup of Myeloproliferative neoplasms (FIM) study. Haematologica. 2018 Mar;103(3):438-446. doi: 10.3324/haematol.2017.181297. Epub 2017 Dec 7. PMID 29217781
- [Result] Mahe K, Delluc A, Chauveau A, Castellant P, Mottier D, Dalbies F, Berthou C, Guillerm G, Lippert E, Ianotto JC. Incidence and impact of atrial arrhythmias on thrombotic events in MPNs. Ann Hematol. 2018 Jan;97(1):101-107. doi: 10.1007/s00277-017-3164-x. Epub 2017 Nov 21. PMID 29164292
- [Result] Ianotto JC, Couturier MA, Galinat H, Mottier D, Berthou C, Guillerm G, Lippert E, Delluc A. Administration of direct oral anticoagulants in patients with myeloproliferative neoplasms. Int J Hematol. 2017 Oct;106(4):517-521. doi: 10.1007/s12185-017-2282-5. Epub 2017 Jun 16. PMID 28623609
- [Result] Le Clech L, Sakka M, Meskar A, Kerspern H, Eveillard JR, Berthou C, Buors C, Lippert E, Guillerm G, Quintin-Roue I, Carre JL, Ianotto JC. The presence of monoclonal gammopathy in Ph-negative myeloproliferative neoplasms is associated with a detrimental effect on outcomes. Leuk Lymphoma. 2017 Nov;58(11):2582-2587. doi: 10.1080/10428194.2017.1312380. Epub 2017 May 9. PMID 28482711
- [Result] Le Gall-Ianotto C, Brenaut E, Gouillou M, Lacut K, Nowak E, Tempescul A, Berthou C, Ugo V, Carre JL, Misery L, Ianotto JC. Clinical characteristics of aquagenic pruritus in patients with myeloproliferative neoplasms. Br J Dermatol. 2017 Jan;176(1):255-258. doi: 10.1111/bjd.14809. Epub 2016 Dec 22. No abstract available. PMID 27291777
- [Derived] Gall-Ianotto CL, Civi L, Pan-Petesch B, Herbreteau L, Rio L, Lambert WC, Misery L, Lippert E, Ianotto JC. Ruxolitinib and Hydroxycarbamide Are the Most Efficient Drugs to Reduce Aquagenic Pruritus Intensity in a Real-Word Cohort of Patients With Myeloproliferative Neoplasms. EJHaem. 2025 Dec 11;6(6):e70197. doi: 10.1002/jha2.70197. eCollection 2025 Dec. PMID 41393215